CLINICAL TRIAL: NCT06883227
Title: Investigating Health Impacts of Exposure to Harmful Algal Blooms
Status: Recruiting | Type: Observational
Sponsor: Roskamp Institute Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: RI-ET-001
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Red Tide; Neurologic Disorder; Florida
Keywords: Brain fog; Red Tide; respiratory; coughing; neurotoxin; beach; florida
MeSH Terms: conditions — Nervous System Diseases; Mental Fatigue; Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Main Study: All subjects will be asked to complete four in-person visits where the goal is for two visits to take place during the K. brevis bloom period and the other two visits will be when there is no K. brevis bloom ("not present" range according to the FWC K. brevis cell counts).
- Sub-Study: Sponsor will enroll 45 randomly selected participants from the main cohort of participants who met the inclusion/exclusion criteria and agreed to take part in the PK sub-study. The only additional exclusion criteria will be pregnancy at the time of PK study. Participants will be asked to take part in the sub-study after their first visit where there was no bloom present. Participants in the relevant locations (areas in which there is red tide bloom present) will be contacted to initiate the PK studies, and data from their prior visit (when there was no red tide bloom present) will represent their baseline data (D0).

SUMMARY:
The goals of this project are to study the biological effects of environmental toxins (ET), in particular aquatic toxins such as brevetoxins (PbTx) and microcystin or their metabolites. This study is designed to examine the effects of the body from harmful algae blooms (HAB) as well as possibility of an association between exposure to the marine toxin, brevetoxin (PbTx), which is released from K. brevis during the red tide bloom, and the prevalence of neurological illnesses.

DETAILED DESCRIPTION:
Exposure to environmental toxins present in local waters, such as brevetoxins released by Karenia brevis (K. brevis) or microcystin produced by cyanobacteria, is known to cause skin and eye irritation, gastrointestinal and respiratory distress. The ingestion of high levels of brevetoxins from eating contaminated shellfish can result in Neurotoxic Shellfish Poisoning (NSP), an acute gastroenteritis with accompanying neurologic symptoms. People are often exposed by direct skin contact with contaminated waters, drinking contaminated water, breathing in airborne droplets of the toxins, or eating contaminated shellfish. This condition usually resolves itself within 3 days as the brevetoxins are excreted from the body. Aerosolized brevetoxins are also known to cause a reversible upper respiratory syndrome, characterized by coughing, sneezing, and feelings of irritation to the airways. Once the exposure to the brevetoxin-laden air has ceased, symptoms usually go away within 15 minutes.

The main objective of this study is to determine if exposure to marine or similar environmental toxins can adversely affect CNS health, immune system, respiratory system and other biological processes which contribute to long-term cognitive dysfunction or illnesses in individuals exposed to these toxins.

Sponsor will be examining whether general health signs and symptoms that are reported are as associated with the exposure to harmful algal bloom toxins. Known symptoms of exposure to harmful algae bloom/red tide /shellfish include the following: Skin and eye irritation, gastrointestinal and respiratory distress, acute gastroenteritis with accompanying neurologic symptoms, respiratory distress, such as reversible upper respiratory syndrome with symptoms of coughing, sneezing, and feelings of irritation to the airways.

ELIGIBILITY:
Inclusion Criteria:

1. Subject should be able to provide written informed consent.
2. Adult aged 18 or older.
3. Resident (temporary or permanent) of one of the following five southwest Florida counties (Lee, Collier, Charlotte, Sarasota, or Manatee).
4. Any race or ethnicity.
5. Willing to return for at least a total of four study visits and participate in all required procedures for the duration of the study.

Exclusion Criteria:

1. Inability to speak or write in English.
2. Any medical condition for which the study investigator believes enrollment is medically inappropriate.
3. Unwilling/unable to provide biological samples or poor venous access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who have been likely exposed to marine toxins (based on the areas that they frequent) as well as individuals who are unlikely to have been exposed will be recruited. Also, residents (temporary or permanent) of one of the following five southwest Florida counties (Lee, Collier, Charlotte, Sarasota, or Manatee).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2029-10-14 (Estimated); Study Completion 2030-10-14 (Estimated)

PRIMARY OUTCOMES:
Examination of marine or similar environmental toxins short-term and long-term adverse effects on central nervous system (CNS) health, immune system, respiratory health and other biological effects induced by aquatic environmental or related toxins. | 4 years
  The Investigators want to examine the effects of the body from harmful algae blooms (HAB) as well as possibility of an association between exposure to the marine toxin, brevetoxin (PbTx), which is released from K. brevis during the red tide bloom, and the prevalence of neurological illnesses. Height and weight will be combined to assess BMI (BMI = weight (lb) ÷ height2 (inches))

CONTACTS AND LOCATIONS:
Overall Officials: Laila Abdullah Principal Investigator, Ph.D, Principal Investigator — The Roskamp Institute
Locations (1):
- The Roskamp Institute, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No